CLINICAL TRIAL: NCT02149264
Title: A Phase 3, Open-Label, Non-Randomized, Clinical Trial to Evaluate the Efficacy and Safety of FE 999303 (Testosterone Gel) in Adult Hypogonadal Males
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Testosterone Gel in Adult Hypogonadal Males
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000127
Record Dates: First submitted 2014-05-19; First posted 2014-05-29 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Adult Male Hypogonadism
MeSH Terms: conditions — Eunuchism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone gel (FE 999303) (Experimental): Subjects received at least one dose of testosterone gel (23 mg), which was further titrated, if needed (upto three doses [69 mg]), based on serum testosterone concentrations. Testosterone gel was delivered using an applicator to the contralateral shoulder/upper arm.
  Interventions: Drug: Testosterone gel (FE 999303)

INTERVENTIONS:
Drug: Testosterone gel (FE 999303)

SUMMARY:
This is a phase 3, open-label, non-randomized, clinical trial to evaluate the efficacy and safety of FE 999303 (Testosterone gel) in adult hypogonadal males.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18-75 years of age
* Two fasting serum testosterone levels <300 ng/dL

Exclusion Criteria:

* Previous use of the study drug
* History of prostate or breast cancer
* Prostate-Specific Antigen (PSA) ≥3 ng/mL
* Subject is sexually active and not willing to use adequate contraception

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (22):
- United States (22):
  - Investigational site, Anniston, Alabama
  - Investigational site, Huntsville, Alabama
  - Investigational site, Newport Beach, California
  - Investigational site, Denver, Colorado
  - Investigational site, New Haven, Connecticut
  - Investigational site, Aventura, Florida
  - Investigational site, Clearwater, Florida
  - Investigational site, Mishawaka, Indiana
  - Investigational site, Watertown, Massachusetts
  - Investigational site, Troy, Michigan
  - Investigational site, Edison, New Jersey
  - Investigational site, Lawrence, New Jersey
  - Investigational site, Garden City, New York
  - Investigational site, New York, New York
  - Investigational site, Poughkeepsie, New York
  - Investigational site, Purchase, New York
  - Investigational site, Bala-Cynwyd, Pennsylvania
  - Investigational site, Warwick, Rhode Island
  - Investigational site, Mt. Pleasant, South Carolina
  - Investigational site, Nashville, Tennessee
  - Investigational site, Webster, Texas
  - Investigational site, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 23 study sites in the United States.
Pre-assignment Details: Of the 940 screened subjects, 160 subjects were eligible to be enrolled into the study.
Groups:
- Testosterone Gel (FE 999303): Subjects received at least one dose of testosterone gel (23 mg), which was further titrated, if needed (up to three doses [69 mg]), based on serum testosterone concentrations. Testosterone gel was delivered using an applicator to the contralateral shoulder/upper arm.
Period: Overall Study
Arm/Group | Testosterone Gel (FE 999303)
Started | 159 (Of the 160 enrolled subjects, one discontinued before receiving treatment.)
Completed | 139
Not Completed | 20
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 7
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population consists of all subjects who received at least one dose of investigational medicinal product (IMP).
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 138
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 137
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 123
  More than one race | 2
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: inches] | 69.8 (2.5)
Weight [Mean (Standard Deviation); unit: lbs] | 213.2 (28.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (3.2)
Total International Index of Erectile Function Score - All Domains [Mean (Standard Deviation); unit: units on a scale] — IIEF questionnaire have 15 questions (Q) divided into 5 domains-
  1. Erectile function (6 items, Q 1-5 and 15) (Score range: 1-30)
  2. Orgasmic function (2 items, Q 9-10) (Score range: 0-10)
  3. Sexual desire (2 items, Q 11-12) (Score range: 2-10)
  4. Intercourse satisfaction (3 items, Q 6-8) (Score range: 0-15)
  5. Overall satisfaction (2 items, Q 13-14) (Score range: 2-10)
  Total score was calculated by summing up scores of each domain and ranged from 5-75. Low score indicates severe dysfunction and a high score indicates no dysfunction in sexual function.
  units on a scale | 36.3 (18.7)
Multidimensional Assessment of Fatigue [Mean (Standard Deviation); unit: units on a scale] — The MAF have 16 questions (Q) divided into 4 domains:
  1. Severity (Q 1-2) (Score range [SR]: 2-20)
  2. Distress (Q 3) (SR: 1-10)
  3. Degree of interference in activities of daily living (Q 4-14) (SR: 11-110)
  4. Timing (Q 15-16) (SR: 5-20)
  First 14 Q are scored from 1-10. Questions 15-16 are scored from 1-4 and converted to 1-10 scale by multiplying each score by 2.5. Lower score in each domain indicates improvement in fatigue.
  GFI was calculated by summing up scores of Q 1, 2, 3, average of 4-14, and revised score of 15. The GFI ranged from 1 (no fatigue) to 50 (severe fatigue).
  units on a scale
    Severity domain | 12.0 (4.9)
    Distress domain | 5.1 (2.6)
    Degree of interference domain | 47.7 (22.9)
    Timing domain | 13.0 (3.0)
    Global Fatigue Index (GFI) | 27.5 (11.1)
Short Form -12 (SF-12) Health survey [Mean (Standard Deviation); unit: units on a scale] — Data collected from the SF-12 questionnaire, based on the norm-based scores is used to assess improvement in the psychometrically-based physical component summary (PCS) and mental component summary (MCS). Both PCS and MCS contains four sub-domains (A total of 12 questions).
  PCS and MCS composite scores are computed using the scores of the 12 questions and range from 0-100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Positive change from baseline indicates improvement in physical and mental health.
  units on a scale
    Physical Component Summary | 48.4 (8.8)
    Mental Component Summary | 43.7 (11.0)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Whose Average Concentration (Cave(0-24)) Serum Total Testosterone Levels Are ≥300 and ≤1050 ng/dL
Description: The data were presented using descriptive statistics. The 95% confidence interval (CI) of the proportion (response) was estimated using the normal approximation to the binomial distribution. The study was considered to have met its efficacy criteria if the percentage was ≥ 75% and the lower bound of the 95% CI was ≥ 65%.
Time Frame: At Day 90
Population: Full Analysis Set (FAS) population was used and included subjects who had sufficient pharmacokinetic data to determine a Cave(0-24) on Days 14, 35, 56, or 90, or discontinued the study early due to medical or safety reasons.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 155
percentage of subjects | 76.1 [69.4 to 82.8]

2. Secondary Outcome: The Percentage of Subjects Whose Cave(0-24) Serum Total Testosterone Levels Are ≥300 and ≤1050 ng/dL
Description: The data were presented using descriptive statistics. No statistical analysis was performed.
Time Frame: At 14, 35 and 56
Population: FAS population was used and included subjects who had sufficient pharmacokinetic data to determine a Cave(0-24) on Days 14, 35, 56, or 90, or discontinued the study early due to medical or safety reasons.
Measure: Number; unit: percentage of subjects
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 155
percentage of subjects
  Day 14 | 29.1
  Day 35 | 58.2
  Day 56 | 71.2

3. Secondary Outcome: Change From Baseline in International Index of Erectile Function (IIEF) Score
Description: Data collected from the five domains of sexual functions were summarized by descriptive statistics. The domains were:
  1. Erectile function (6 items, questions 1-5 and 15) (Score range:1-30)
  2. Orgasmic function (2 items, questions 9-10) (Score range: 0-10)
  3. Sexual desire (2 items, questions 11-12) (Score range: 2-10)
  4. Intercourse satisfaction (3 items, questions 6-8) (Score range: 0-15)
  5. Overall satisfaction (2 items, questions 13-14) (Score range: 2-10)
  A score of 0-5 is awarded to questions 1 to 10 and a score of 1-5 is awarded to questions 11 to 15. Total score was calculated by summing up scores of each domain and ranged from 5 to 75. Low score indicates severe dysfunction and a high score indicates no dysfunction in sexual function.
Time Frame: At Days 35 and 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 155
units on a scale
  Day 35 | 8.4 (13.2)
  Day 90 | 14.4 (16.9)

4. Secondary Outcome: Change From Baseline in Multidimensional Assessment of Fatigue (MAF) Score
Description: The MAF contains four sub-domains:
  1. Severity (2 items, questions 1-2) (Score range: 2-20)
  2. Distress (1 item, question 3) (Score range: 1-10)
  3. Degree of interference in activities of daily living (11 items, questions 4-14) (Score range: 11-110)
  4. Timing (2 items, questions 15-16) (Score range: 5-20)
  A score of 1-10 is awarded to each of the 14 questions across the 3 domains. The timing domain (categorical in nature) are scored from 1-4. The scores are converted to 1-10 scale by multiplying each score by 2.5. Lower score in each domain indicates improvement in fatigue.
  To calculate GFI : Score of question 15 is converted to a 0-10 scale by multiplying each score by 2.5 and then sum questions 1, 2, 3, average of 4-14, and newly scored question 15. A score of zero is assigned to question 2-16, if patient select 'no fatigue' to question 1. Question 16 is not included in GFI calculation. The GFI ranged from 1 (no fatigue) to 50 (severe fatigue).
Time Frame: At Days 35 and 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 155
units on a scale
  Severity domain score at Day 35 | -3.6 (4.8)
  Distress domain score at Day 35 | -1.7 (2.6)
  Degree of interference domain score at Day 35 | -13.6 (24.1)
  Timing domain score at Day 35 | -2.6 (3.3)
  GFI score at Day 35 | -8.3 (10.1)
  Severity domain score at Day 90 | -5.2 (4.9)
  Distress domain score at Day 90 | -2.2 (2.5)
  Degree of interference domain score at Day 90 | -16.7 (24.5)
  Timing domain score at Day 90 | -3.0 (3.4)
  GFI score at Day 90 | -12.0 (11.1)

5. Secondary Outcome: Change From Baseline in Short Form-12 Health Survey (SF-12) Score
Description: Data collected from the SF-12 questionnaire, based on the norm-based scores was used to assess improvement in the psychometrically-based physical component summary (PCS) and mental component summary (MCS). Both PCS and MCS contained four sub-domains:
  PCS:
  1. Physical Functioning (2 items, questions 2-3)
  2. Role-Physical (2 items, questions 4-5)
  3. Bodily Pain (1 item, question 8)
  4. General Health (1 item, question 1)
  MCS:
  1. Vitality (1 item, question 10)
  2. Social Functioning (1 item, question 12)
  3. Role-Emotional (2 items, questions 6-7)
  4. Mental Health (2 items, questions 9 and 11)
  PCS and MCS composite scores are computed using the scores of the 12 questions and range from 0-100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Positive change from baseline indicated improvement in physical and mental health.
Time Frame: At Days 35 and 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 155
units on a scale
  PCS Day 35 | 1.2 (7.0)
  PCS Day 90 | 1.8 (7.1)
  MCS Day 35 | 6.3 (9.5)
  MCS Day 90 | 6.5 (10.1)

6. Secondary Outcome: Pharmacokinetic Parameter - Average Concentration (Cave) for Total Testosterone and Dihydrotestosterone
Description: A validated high pressure liquid chromatography with tandem mass spectrometry detection (LC/MS/MS) method was used to determine the levels of total testosterone and dihydrotestosterone.
Time Frame: Samples collected at pre-dose, 2, 4, 6, 8 & 24 hours post-dose on Days 14, 35 & 56, and at pre-dose, 2, 4, 6, 8, 10, 12, 18 & 24 hours post-dose on Day 90
Population: FAS population was used and included subjects who had sufficient pharmacokinetic data to determine a Cave(0-24) on Days 14, 35, 56, or 90, or discontinued the study early due to medical or safety reasons. Number of subjects was less than 155 in some group(s) as parameter could not be calculated due to missing concentrations for that time-point.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 155
ng/dL
  Total testosterone on Day 14 at 23 mg dose: number analyzed (Participants) | 151
  Total testosterone on Day 14 at 23 mg dose | 268 (80)
  Total testosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Total testosterone on Day 35 at 23 mg dose | 359 (116)
  Total testosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 127
  Total testosterone on Day 35 at 46 mg dose | 361 (152)
  Total testosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Total testosterone on Day 56 at 23 mg dose | 278 (73)
  Total testosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Total testosterone on Day 56 at 46 mg dose | 429 (127)
  Total testosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 73
  Total testosterone on Day 56 at 69 mg dose | 464 (271)
  Total testosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Total testosterone on Day 90 at 23 mg dose | 368 (121)
  Total testosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Total testosterone on Day 90 at 46 mg dose | 506 (207)
  Total testosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Total testosterone on Day 90 at 69 mg dose | 438 (164)
  Dihydrotestosterone on Day 14 at 23 mg dose: number analyzed (Participants) | 150
  Dihydrotestosterone on Day 14 at 23 mg dose | 40.9 (18.8)
  Dihydrotestosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Dihydrotestosterone on Day 35 at 23 mg dose | 56.3 (18.0)
  Dihydrotestosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 127
  Dihydrotestosterone on Day 35 at 46 mg dose | 63.1 (29.9)
  Dihydrotestosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Dihydrotestosterone on Day 56 at 23 mg dose | 44.2 (11.1)
  Dihydrotestosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Dihydrotestosterone on Day 56 at 46 mg dose | 78.7 (32.8)
  Dihydrotestosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 73
  Dihydrotestosterone on Day 56 at 69 mg dose | 75.2 (43.3)
  Dihydrotestosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Dihydrotestosterone on Day 90 at 23 mg dose | 65.9 (24.1)
  Dihydrotestosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Dihydrotestosterone on Day 90 at 46 mg dose | 91.2 (38.9)
  Dihydrotestosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Dihydrotestosterone on Day 90 at 69 mg dose | 77.7 (39.7)

7. Secondary Outcome: Pharmacokinetic Parameter - Area Under the Concentration-time Curve (AUCτ) for Total Testosterone and Dihydrotestosterone
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone and dihydrotestosterone.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 155
ng*hr/dL
  Total testosterone on Day 14 at 23 mg dose: number analyzed (Participants) | 151
  Total testosterone on Day 14 at 23 mg dose | 6431 (1938)
  Total testosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Total testosterone on Day 35 at 23 mg dose | 8552 (2800)
  Total testosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 127
  Total testosterone on Day 35 at 46 mg dose | 8665 (3664)
  Total testosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Total testosterone on Day 56 at 23 mg dose | 6624 (1765)
  Total testosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Total testosterone on Day 56 at 46 mg dose | 10320 (3042)
  Total testosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 73
  Total testosterone on Day 56 at 69 mg dose | 11152 (6507)
  Total testosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Total testosterone on Day 90 at 23 mg dose | 8831 (2829)
  Total testosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Total testosterone on Day 90 at 46 mg dose | 12245 (5010)
  Total testosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Total testosterone on Day 90 at 69 mg dose | 10590 (3979)
  Dihydrotestosterone on Day 14 at 23 mg dose: number analyzed (Participants) | 150
  Dihydrotestosterone on Day 14 at 23 mg dose | 980 (452)
  Dihydrotestosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Dihydrotestosterone on Day 35 at 23 mg dose | 1343 (435)
  Dihydrotestosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 127
  Dihydrotestosterone on Day 35 at 46 mg dose | 1515 (719)
  Dihydrotestosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Dihydrotestosterone on Day 56 at 23 mg dose | 1057 (270)
  Dihydrotestosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Dihydrotestosterone on Day 56 at 46 mg dose | 1893 (797)
  Dihydrotestosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 73
  Dihydrotestosterone on Day 56 at 69 mg dose | 1811 (1046)
  Dihydrotestosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Dihydrotestosterone on Day 90 at 23 mg dose | 1579 (560)
  Dihydrotestosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Dihydrotestosterone on Day 90 at 46 mg dose | 2210 (956)
  Dihydrotestosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Dihydrotestosterone on Day 90 at 69 mg dose | 1876 (956)

8. Secondary Outcome: Pharmacokinetic Parameter - Time at Which the Maximum Concentration Occurs (Tmax) for Total Testosterone and Dihydrotestosterone
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone and dihydrotestosterone.
Time Frame: as for outcome 6
Population: FAS population was used and included subjects who had sufficient pharmacokinetic data to determine a Cave(0-24) on Days 14, 35, 56, or 90, or discontinued the study early due to medical or safety reasons. Of 155 subjects, one subject discontinued due to adverse event after Day 14 visit and not included in the analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 154
hr
  Total testosterone on Day 14 at 23 mg dose | 2.04 [0.0 to 24.9]
  Total testosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Total testosterone on Day 35 at 23 mg dose | 2.15 [0.0 to 23.8]
  Total testosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 128
  Total testosterone on Day 35 at 46 mg dose | 2.00 [0.0 to 24.9]
  Total testosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Total testosterone on Day 56 at 23 mg dose | 2.00 [1.75 to 4.05]
  Total testosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Total testosterone on Day 56 at 46 mg dose | 2.08 [0.0 to 24.3]
  Total testosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 75
  Total testosterone on Day 56 at 69 mg dose | 2.00 [0.0 to 24.1]
  Total testosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Total testosterone on Day 90 at 23 mg dose | 4.02 [2.00 to 6.00]
  Total testosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Total testosterone on Day 90 at 46 mg dose | 2.02 [1.75 to 25.4]
  Total testosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Total testosterone on Day 90 at 69 mg dose | 2.08 [0.0 to 24.8]
  Dihydrotestosterone on Day 14 at 23 mg dose | 3.97 [0.0 to 24.6]
  Dihydrotestosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Dihydrotestosterone on Day 35 at 23 mg dose | 3.04 [0.0 to 7.97]
  Dihydrotestosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 128
  Dihydrotestosterone on Day 35 at 46 mg dose | 2.94 [0.0 to 25.1]
  Dihydrotestosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Dihydrotestosterone on Day 56 at 23 mg dose | 2.00 [1.75 to 4.17]
  Dihydrotestosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Dihydrotestosterone on Day 56 at 46 mg dose | 2.08 [0.0 to 24.5]
  Dihydrotestosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 75
  Dihydrotestosterone on Day 56 at 69 mg dose | 3.87 [0.0 to 24.8]
  Dihydrotestosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Dihydrotestosterone on Day 90 at 23 mg dose | 4.12 [0.0 to 23.5]
  Dihydrotestosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Dihydrotestosterone on Day 90 at 46 mg dose | 3.75 [0.0 to 25.4]
  Dihydrotestosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Dihydrotestosterone on Day 90 at 69 mg dose | 3.95 [0.0 to 24.9]

9. Secondary Outcome: Pharmacokinetic Parameter - Maximum Concentration Observed (Cmax) for Total Testosterone and Dihydrotestosterone
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone and dihydrotestosterone.
Time Frame: as for outcome 6
Population: FAS population was used and included subjects who had sufficient pharmacokinetic data to determine a Cave(0-24) on Days 14, 35, 56, or 90, or discontinued the study early due to medical or safety reasons. Of 155 subjects, one subject discontinued due to an adverse event after Day 14 visit and not included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 154
ng/dL
  Total testosterone on Day 14 at 23 mg dose | 435 (195)
  Total testosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Total testosterone on Day 35 at 23 mg dose | 642 (238)
  Total testosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 128
  Total testosterone on Day 35 at 46 mg dose | 732 (387)
  Total testosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Total testosterone on Day 56 at 23 mg dose | 637 (300)
  Total testosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Total testosterone on Day 56 at 46 mg dose | 890 (424)
  Total testosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 75
  Total testosterone on Day 56 at 69 mg dose | 987 (652)
  Total testosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Total testosterone on Day 90 at 23 mg dose | 721 (254)
  Total testosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Total testosterone on Day 90 at 46 mg dose | 1228 (640)
  Total testosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Total testosterone on Day 90 at 69 mg dose | 1099 (595)
  Dihydrotestosterone on Day 14 at 23 mg dose | 56.5 (26.9)
  Dihydrotestosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Dihydrotestosterone on Day 35 at 23 mg dose | 79.2 (26.0)
  Dihydrotestosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 128
  Dihydrotestosterone on Day 35 at 46 mg dose | 91.5 (43.3)
  Dihydrotestosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Dihydrotestosterone on Day 56 at 23 mg dose | 68.6 (19.0)
  Dihydrotestosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Dihydrotestosterone on Day 56 at 46 mg dose | 113 (62)
  Dihydrotestosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 75
  Dihydrotestosterone on Day 56 at 69 mg dose | 106 (57)
  Dihydrotestosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Dihydrotestosterone on Day 90 at 23 mg dose | 91.4 (34.8)
  Dihydrotestosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Dihydrotestosterone on Day 90 at 46 mg dose | 138 (66)
  Dihydrotestosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Dihydrotestosterone on Day 90 at 69 mg dose | 118 (55)

10. Secondary Outcome: Pharmacokinetic Parameter - Minimum Concentration Observed (Cmin) for Total Testosterone and Dihydrotestosterone
Description: A validated LC/MS/MS method was used to determine the levels of total testosterone and dihydrotestosterone.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 154
ng/dL
  Total testosterone on Day 14 at 23 mg dose | 194 (64)
  Total testosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Total testosterone on Day 35 at 23 mg dose | 203 (74)
  Total testosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 128
  Total testosterone on Day 35 at 46 mg dose | 216 (93)
  Total testosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Total testosterone on Day 56 at 23 mg dose | 175 (49)
  Total testosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Total testosterone on Day 56 at 46 mg dose | 262 (115)
  Total testosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 75
  Total testosterone on Day 56 at 69 mg dose | 261 (200)
  Total testosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Total testosterone on Day 90 at 23 mg dose | 191 (49)
  Total testosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Total testosterone on Day 90 at 46 mg dose | 277 (140)
  Total testosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Total testosterone on Day 90 at 69 mg dose | 229 (82)
  Dihydrotestosterone on Day 14 at 23 mg dose | 30.7 (15.6)
  Dihydrotestosterone on Day 35 at 23 mg dose: number analyzed (Participants) | 18
  Dihydrotestosterone on Day 35 at 23 mg dose | 41.0 (12.7)
  Dihydrotestosterone on Day 35 at 46 mg dose: number analyzed (Participants) | 128
  Dihydrotestosterone on Day 35 at 46 mg dose | 43.9 (24.7)
  Dihydrotestosterone on Day 56 at 23 mg dose: number analyzed (Participants) | 8
  Dihydrotestosterone on Day 56 at 23 mg dose | 33.2 (9.6)
  Dihydrotestosterone on Day 56 at 46 mg dose: number analyzed (Participants) | 59
  Dihydrotestosterone on Day 56 at 46 mg dose | 58.0 (26.7)
  Dihydrotestosterone on Day 56 at 69 mg dose: number analyzed (Participants) | 75
  Dihydrotestosterone on Day 56 at 69 mg dose | 52.9 (32.3)
  Dihydrotestosterone on Day 90 at 23 mg dose: number analyzed (Participants) | 5
  Dihydrotestosterone on Day 90 at 23 mg dose | 45.1 (21.0)
  Dihydrotestosterone on Day 90 at 46 mg dose: number analyzed (Participants) | 45
  Dihydrotestosterone on Day 90 at 46 mg dose | 62.5 (26.4)
  Dihydrotestosterone on Day 90 at 69 mg dose: number analyzed (Participants) | 89
  Dihydrotestosterone on Day 90 at 69 mg dose | 53.1 (29.7)

ADVERSE EVENTS:
Time Frame: Overall study period (From Day 1 to Day 120 [last visit])
Description: Adverse event occurring after start of study drug administration and within the time of residual drug effect (5 days), or a pre-treatment adverse event or pre-existing medical condition that worsened in intensity after treatment with the study drug and within the time of residual drug effect, are presented for the safety analysis set.
Arm/Group | Testosterone Gel (FE 999303)
Serious Adverse Events (participants affected / at risk) | 5/159
Other Adverse Events (participants affected / at risk) | 54/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Gel (FE 999303) (N=159)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone Gel (FE 999303) (N=159)
Hydrocele (Congenital, familial and genetic disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Application site dermatitis (General disorders) | 1
Application site erythema (General disorders) | 4
Application site pruritus (General disorders) | 1
Application site rash (General disorders) | 3
Cyst (General disorders) | 1
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Sluggishness (General disorders) | 1
Bronchitis (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Perineal abscess (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 2
Blood pressure increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 3
Gamma-glutamyl transferase increased (Investigations) | 2
Glycosylated haemoglobin increased (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 2
Weight increased (Investigations) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hyposmia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Breast tenderness (Reproductive system and breast disorders) | 1
Epididymitis (Reproductive system and breast disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 2
Nipple pain (Reproductive system and breast disorders) | 1
Prostatic pain (Reproductive system and breast disorders) | 1
Testicular atrophy (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.